CLINICAL TRIAL: NCT01546337
Title: Search for Predictive Markers of Efficacy of Epoetin Beta (NEORECORMON) in the Treatment of Anemia in Patients With Non-myeloid Malignancies Receiving Chemotherapy or Myelodysplastic Syndrome
Brief Title: Search for Predictive Markers of Efficacy of ESAs in Patients With Non-myeloid Malignancies or Myelodysplastic Syndrome
Acronym: EPO
Status: Terminated | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCTIRS908111
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Myelodysplastic Syndromes; Anemia; Hemopathies
Keywords: anemia; non-myeloid haemopathy; myelodysplastic syndrome; Erythropoiesis stimulating agents; predictive markers
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anemia is common among cancer patients and the treatment of choice is now Erythropoiesis-Stimulating Agents (ESAs). However, some patients do not respond to treatment. The purpose of this study is to evaluate the predictive value of endogenous erythropoietin rate on the response to erythropoietin beta. First, by confirming the predictive value of endogenous erythropoietin observed / predicted ratio on this response. Then if it is confirmed by establishing the optimal value of this ratio.

DETAILED DESCRIPTION:
Anemia is common among cancer patients and the treatment of choice is now Erythropoiesis-Stimulating Agents (ESAs). However, some patients do not respond to treatment. Thus, only 50-60% of patients with multiple myeloma or non-Hodgkin lymphoma respond to ESAs. The purpose of this study is to evaluate the predictive value of endogenous erythropoietin rate on the response to erythropoietin beta. First, by confirming the predictive value of endogenous erythropoietin observed / predicted ratio on this response. Then if it is confirmed by establishing the optimal value of this ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* patients with non-myeloid haemopathy receiving chemotherapy or myelodysplastic syndrome
* indication of ESAs therapy with Hb < 11g/dl

Exclusion Criteria:

* uncontrolled hypertension
* anemia due to deficiency
* pregnant and lactating women
* patient who received treatment with erythropoiesis-activating factors in the two months preceding inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-myeloid haemopathy or Myelodysplastic Syndromes patients with anemia, who needs ESAs treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
response to erythropoietin | 12 weeks
  * Complete response : increase of 2g/dl of erythropoietin rate or stopping of transfusion requirements.
  * Partial response : increase of 1 to 2g/dl rate of erythropoietin or 50% reduction of transfusion requirements.

SECONDARY OUTCOMES:
endogenous erythropoietin rate | Within 8 days before inclusion
hemoglobin rate | Weeks 0,4,8 and 12
  Weeks 0 = first ESAs injection
Number of transfusions during the duration of the study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Escoffre-Barbe Martine, MD, Principal Investigator — Rennes University Hospital; Laviolle Bruno, MD, Study Chair — Rennes University Hospital
Locations (5):
- France (5):
  - Laval Hospital, Laval
  - Rennes University Hospital, Rennes
  - Yves Le Foll Hospital, Saint-Brieuc
  - Saint-Malo Hospital, St-Malo
  - Bretagne Atlantic Hospital, Vannes